CLINICAL TRIAL: NCT01562691
Title: Comparison of Nasal Packing Methods:Nasal Packing Was Done With Nasopore@, Airway-integrated Nasopore@ and Airway-integrated Vaseline Gauze
Brief Title: Effect of Airway Integrated Nasal Packing With Different Material
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Yung-Song Lin, Chairman of department of Otolaryngology, Chi Mei Medical Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CMH-09706-001
Record Dates: First submitted 2012-03-21; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Respiratory Complications; Pain, Postoperative.
Keywords: nasal packing; nasal airway; septoplasty; oxygen saturation; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nasopore only (Experimental): Packing using nasopore without airway integrated
  Interventions: Procedure: Nasopore
- nasopore with airway integrated (Active Comparator): packing using airway integrated nasopore
  Interventions: Procedure: airway integrated Nasopore
- airway-integrated Vaseline gauze (Active Comparator): Nasal packing using airway-integrated Vaseline gauze
  Interventions: Procedure: airway-integrated Vaseline gauze

INTERVENTIONS:
Procedure: Nasopore — Bilateral nasal packing using Nasopore without airway integrated
  Arms: Nasopore only
Procedure: airway integrated Nasopore — post nasoseptoplasty with nasal packing using airway integrated Nasopore
  Arms: nasopore with airway integrated
Procedure: airway-integrated Vaseline gauze — post nasal septoplasty with packing using airway-integrated Vaseline gauze
  Arms: airway-integrated Vaseline gauze

SUMMARY:
The purpose of this study is to determine the effect of integrated airway in nasal packing material foe patients receiving nasal septoplasty surgery.

DETAILED DESCRIPTION:
Nasal packing with integrated airway had been claimed to improve body oxygenation following septal surgery. This randomized control study examined the effect of airway integrated with nasal packing, in terms of its improvement on oxygen saturation. Sixty patients with septal deviation and hypertrophic turbinate were randomized into three groups. Group 1 patients were packed with only nasopore@ after surgery. Nasopore@ with integrated airway was used for group 2 patients; and Vaseline gauze integrated with airway for group 3 patients. Hemodynamic parameters were sequentially checked. Nasal pain sensation was recorded using visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent septoplasty for septal deviation and chronic hypertrophic rhinitis

Exclusion Criteria:

* patients with comorbidities of coronary heart disease, arrhythmia, chronic obstructive lung diseases, and with past history of any nasal surgery were excluded.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
oxyhemoglobin saturation by pulse oximetry, SpO2 | SpO2 was measured 30 minutes before operation,
  SpO2 was measured 30 minutes before operation using O2 saturation monitor.
change of SpO2 from baseline to 4 hours post-operation | records of the SpO2 at 4 hours post-operation
  records of the SpO2 at 4 hours post-operation
change of the SpO2 from baseline to 6 hours post-operation | records of the SpO2 at 6 hours post-operation
  records of the SpO2 at 6 hours post-operation
change of the SpO2 from baseline to 12 hours post-operation | records of the SpO2 at 12 hours post-operation
  records of the SpO2 at 12 hours post-operation
change of the SpO2 from baseline to 18 hours post-operation | records of the SpO2 at 18 hours post-operation
  records of the SpO2 at 18 hours post-operation
change of the SpO2 from baseline to 48 hours post-operation | records of the SpO2 at 48 hours post-operation
  records of the SpO2 at 48 hours post-operation

SECONDARY OUTCOMES:
postoperation pain | record of postoperation pain scale at 2 hous post operation
  record of postoperation pain scale at 2 hours post-operation
change of postoperation pain scale from baseline to 4 hours post-operation | record of postoperation pain scale at 4 hours post-operation
  record of postoperation pain scale at 4 hours post-operation
change of postoperation pain scale from baseline to 6 hours post-operation | Record of postoperation pain scale at 6 hours post-operation
  record of postoperation pain scale at 6 hours post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Song Lin, M.D., Study Chair — Chi Mei Medical Hospital
Locations (1):
- Chi Mei Medical Center, Tainan, Taiwan, Taiwan